CLINICAL TRIAL: NCT00377481
Title: A Randomised, Cross-Over Study to Investigate the Comfort of Injection of Renal Anaemia Patients Receiving Subcutaneous NeoRecormon® Compared to Darbepoetin Alfa.
Brief Title: COMFORT Study: A Crossover Study of NeoRecormon (Epoetin Beta) and Darbepoetin Alfa in Patients With Renal Anemia.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: ML20339
Record Dates: First submitted 2006-09-15; First posted 2006-09-18 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — Darbepoetin alfa; epoetin beta

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: epoetin beta [NeoRecormon]
- 2 (Active Comparator)
  Interventions: Drug: darbepoetin alfa

INTERVENTIONS:
Drug: darbepoetin alfa — 30 micrograms sc weekly (2 doses)
  Arms: 2
Drug: epoetin beta [NeoRecormon] — 6000 IU sc weekly (2 doses)
  Arms: 1

SUMMARY:
This study will assess the comfort of subcutaneous injections of NeoRecormon and darbepoetin alfa (Aranesp) in patients with renal anemia. Eligible patients will be randomized to receive comparable subcutaneous injections of either darbepoetin alfa (30 micrograms) or NeoRecormon (6000IU). They will then be crossed over to the alternative treatment arm for further treatment. After each injection pain will be assessed using the visual analogue scale (VAS) and 6-point verbal rating scale (VRS), and patient preference will be assessed. The anticipated time on study treatment is <3 months, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >18 years of age;
* patients with renal anemia or post-transplant anemia.

Exclusion Criteria:

* poorly controlled hypertension;
* known hypersensitivity to NeoRecormon or darbepoetin alfa.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2006-09; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Local pain due to s.c. injection (by VAS). | After each injection

SECONDARY OUTCOMES:
Patient preference. | At end of study
AEs, vital signs. | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (8):
- Australia (8):
  - Adelaide
  - Gosford
  - Liverpool
  - Melbourne
  - Parkville
  - St Leonards
  - Sydney
  - Woolloongabba

REFERENCES:
- [Derived] Roger SD, Suranyi MG, Walker RG, Disney A, Isbel NM, Kairaitis L, Pollock CA, Brown FG, Chow J, Truman MI, Ulyate KA; COMFORT study group. A randomised, cross-over study comparing injection site pain with subcutaneous epoetin beta and subcutaneous darbepoetin alfa in patients with chronic kidney disease. Curr Med Res Opin. 2008 Aug;24(8):2181-7. doi: 10.1185/03007990802240552. Epub 2008 Jun 18. PMID 18565240